CLINICAL TRIAL: NCT06399042
Title: A Multi-center, Randomized, Double-Blinded, Active Controlled, Phase III Study to Evaluate Efficacy and Safety of SP5M002 Injection Compared With Synovian Injection in Patients With Mild to Moderate Knee Osteoarthritis
Brief Title: Pivotal Study to Evaluate Efficacy and Safety of SP5M002 Inj. as Compared to Synovian Inj. in Patients With Mild to Moderate Knee Osteoarthritis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-HA-003-1
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis
Keywords: Knee osteoarthritis, Intra-articular injection, hexamethylenediamine(HMDA), Cross-linked hyaluronate
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: masking : only blind investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SP5M002 inj (Experimental): SP5M002 inj 3 ml pre-filled syringe into Knee joint cavity of osteoarthritis patients
  Interventions: Device: SP5M002 inj
- Synovian inj (Active Comparator): Synovian inj 3 ml pre-filled syringe into Knee joint cavity of osteoarthritis patients
  Interventions: Device: Synovian inj

INTERVENTIONS:
Device: SP5M002 inj — pre-filled syringe
  Arms: SP5M002 inj
Device: Synovian inj — pre-filled syringe
  Arms: Synovian inj

SUMMARY:
This is a randomized, double-blind, multicenter, Active Controlled, pivotal clinical trial to assess the efficacy and safety of the novel hexamethylenediamine (HMDA) cross-linked hyaluronate intra-articular injection (SP5M002) compared with an active comparator, the 1,4-butanediol diglycidyl ether (BDDE) cross-linked hyaluronate (Synovian) in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged 40 years or older as of the date of written consent
2. Subject with knee osteoarthritis whose X-ray test results within 6 months from the screening or at the screening visit correspond to grades I - III of the Kellgren & Lawrence scale
3. Subject diagnosed with unilateral or bilateral knee osteoarthritis according to the clinical diagnostic criteria of the American College of Rheumatology (ACR) at screening who have knee joint pain and meet three or more of the following conditions

   * Over 50 years of age

     * Less than 30 minutes of morning stiffness ③ Crepitus on active motion ④ Bony tenderness ⑤ Bony enlargement ⑥ No palpable warmth of synovium
4. Weight bearing pain (WBP) of at least one of both knee joints on 100 mm-VAS ≥ 40 mm when measured at screening and baseline [However, if both sides have symptoms, the knee joint with the higher WBP becomes the joint for evaluation, and the selected joint cannot be changed during the study period.]
5. Walk without relying on a walking aid such as a walker or cane (patients who have been using a walking aid every day since 6 months prior to the screening visit can use the walking aid, and must use the walking aid in the same way throughout the study period.)
6. Ability to fully understand and complete the safety and efficacy measurement questionnaire
7. Voluntary decision for participation and provision of written consent to comply with the precautions after hearing and fully understanding the detailed explanation of the purpose, method, and effects of this study

Exclusion Criteria:

1. Body mass index (BMI) ≥ 35 kg/m2 at screening
2. Hip osteoarthritis or osteoarthritis of another joint that is severe enough to preclude evaluation of knee osteoarthritis at the time of screening
3. Having the following diseases that may affect the efficacy and safety evaluation but not being limited to the following

   * Septic arthritis, rheumatoid arthritis, gout, recurrent pseudogout arthritis, trauma that may damage joint cartilage, congenital abnormalities, calcium deposition disease, diabetes, ochronosis, hemochromatosis, acromegaly, Wilson's disease, primary osteochondrosis, genetic diseases (e.g., hyperkinesis), secondary osteoarthritis caused by collagen gene abnormalities, etc.
   * Sudek's atrophy or severe painful diseases such as Paget's disease
4. Infection or skin disease in the joint area that is unsuitable for injection at the time of screening
5. Active or suspected knee joint infection at the time of screening
6. Complete loss of the Patello-femoral joint space
7. Received the following treatments within 14 days of the screening visit (except those who have passed a 14-day wash-out) or scheduled to be administered during the study period

   * Taking medicines containing ingredients such as glucosamine, chondroitin sulfate, and diacerhein
   * Taking herbal medicines and herbal medicines for osteoarthritis
   * Taking anti-inflammatory painkillers, non-steroidal anti-inflammatory drugs (NSAIDs, prescription/non-prescription drugs), etc. (administration of acetaminophen allowed if passing a 3 day wash-out)
   * Taking oral steroids
   * Hospital physical therapy or oriental medicine treatment (cupping, acupuncture, moxibustion, etc.)
8. Intra-articular injection, such as intra-articular corticosteroid, at the injection site within 6 months from the time of screening
9. Systemic use of steroids within 3 months from the time of screening (including inhalants, however, topical application is permitted only on the upper body)
10. Surgical operations such as knee joint replacement, including arthroscopic surgery, at the administration site within 6 months from the time of screening; or expecting surgery within 6 months
11. Moderate or severe joint effusion by Patella tap test at the screening visit
12. History of hypersensitivity to ingredients of the IP or active control drug
13. Antiplatelet agents (excluding aspirin of 300 mg/day or less), heparin, oral anticoagulants (coumarin anticoagulants, thrombin inhibitors, Factor Xa inhibitors, etc.), and thrombolytics must be used during the study
14. Clinically significant abnormalities in liver function (3 times or more than the upper limit of normal for ALT/AST) or abnormalities in renal function (3 times or more than the upper limit of normal for serum creatinine), or severe liver or renal disease at the discretion of the investigator which is judged to have an impact on the effectiveness and safety evaluation of the study
15. The following clinically significant diseases in the past or present

    * Diagnosis of malignancy within 5 years prior to screening or currently
    * Cardiac disorders (myocardial infarction, coronary artery bypass surgery, arrhythmia, and other serious Cardiac disorders, etc.)
    * Uncontrolled hypertension (systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg)
    * Severe endocrine diseases (diabetes insipidus, Cushing's disease, etc.) which is judged to have an impact on the efficacy and safety evaluation of the study
16. Currently pregnant or lactating; or planning to become pregnant/lactating during this study
17. Women of childbearing age who have not undergone sterilization surgery, women less than 1 year after menopause, or men who do not agree to avoid pregnancy or use appropriate contraceptive methods during the study period
18. Planned to participate in another study during the study period or having administered (applied) other investigational product (investigational device) within 3 months prior to the screening visit
19. Difficult to conduct the study as judged by the investigator due to other reasons

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in [Weight-Bearing Pain (WBP)-100mm-visual analogue scale (VAS)] at Week 12 from baseline (visit 2) | 12 weeks
  * Weight Bearing Pain (WBP) - 100mm-visual analogue scale (VAS)
Change in [Weight-Bearing Pain (WBP)-100mm-visual analogue scale (VAS)] at Week 6 from baseline (visit 2) | 6 weeks
  * Weight Bearing Pain (WBP) - 100mm-visual analogue scale (VAS)

SECONDARY OUTCOMES:
Changes in the following at each visit: Weight Bearing pain (WBP) (Weeks 2, 24, and 36) from baseline (Visit 2) | week 2, 24, 36
  Outcome Measurement of Weight Bearing pain(WBP): 100mm-visual analogue scale (VAS)
Changes in the following at each visit: Rest pain (RP) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2,6,12, 24, 36
  Outcome Measurement of Rest pain (RP): 100mm-visual analogue scale (VAS)
Changes in the following at each visit: Night pain (NP) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2,6,12, 24, 36
  Outcome Measurement of Night pain (NP): 100mm-visual analogue scale (VAS)
Changes in the following at each visit: Motion pain (MP) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2,6,12, 24, 36
  Outcome Measurement of Motion pain (MP): 100mm-visual analogue scale (VAS)
Changes in the following at each visit: Patient Global Assessment(PGA) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2,6,12, 24, 36
  Outcome Measurement of Patient Global Assessment(PGA): 100mm-visual analogue scale (VAS)
Changes in the following at each visit: Investigator Global Assessment (IGA) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2,6,12, 24, 36
  Outcome Measurement of Investigator Global Assessment (IGA) : 100mm-visual analogue scale (VAS)
Changes in the following at each visit: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score and individual score evaluation (Pain, function, stiffness) (Weeks 2, 6, 12, 24, and 36) from baseline (Visit 2) | week 2,6,12, 24, 36
  Outcome Measurement of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score and individual score evaluation (Pain, function, stiffness) : WOMAC-Likert Assessment (5-point Likert scale)
Physical assessments at each post-administration visit: Swelling (Weeks 2, 6, 12, 24, and 36) | week 2,6,12, 24, 36
  Outcome Measurement of Swelling : 4-point scale
  *4-point scale: 0(none)/1(mild)/2(moderate)/3(severe)
Physical assessments at each post-administration visit: joint-line tenderness on pressure (Weeks 2, 6, 12, 24, and 36) | week 2,6,12, 24, 36
  Outcome Measurement of joint-line tenderness on pressure : 4-point scale
  *4-point scale: 0(none)/1(mild)/2(moderate)/3(severe)
Physical assessments at each post-administration visit: range of motion (Weeks 2, 6, 12, 24, and 36) | week 2,6,12, 24, 36
  The angle was recorded as is for the range of motion.
Proportion (%) of participants who took rescue medication at each post-administration visit and dose of rescue medication (Weeks 2, 6, 12, 24, and 36) | week 2,6,12, 24, 36
Post-administration response rate A. Proportion at which WBP decreases by at least 20 mm or improves by at least 40% from baseline at the time of evaluation (B section-Description) | week 2,6,12, 24, 36
  *B. Response rate of OMERACT-OARSI (Outcome Measures in Rheumatology-Osteoarthritis Research Society International) I. At least 50% improvement in WOMAC pain or function at the time of evaluation; or at least a 20 point improvement from baseline; or II. meeting 2 of the 3 conditions below
  At least 20% improvement in WOMAC pain, at least a 10 point improvement from each baseline At least 20% improvement in WOMAC function, at least a 10 point improvement from each baseline At least 20% improvement in patient's global assessment (100 mm-VAS) and at least a 10 point improvement from each baseline

OTHER OUTCOMES:
The incidence rate of Pre-treatment AEs | From Week 0 to week 24
The incidence rate of Solicited Local AEs | From Week 0 to week 24
The incidence rate of treatment-emergent adverse event (TEAE) | From Week 0 to week 24
The incidence rate of Serious TEAEs | From Week 0 to week 24
The incidence rate of Serious TEAEs leading to Drug withdrawn | From Week 0 to week 24
The incidence rate of Serious TEAEs leading to Death | From Week 0 to week 24
The incidence rate of abnormal CS at Post-Treatment on Laboratory | From Week 0 to week 24
The incidence rate of abnormal CS at Post-Treatment on Electrocardiogram | From Week 0 to week 24
The incidence rate of abnormal on Physical Examination | From Week 0 to week 24

CONTACTS AND LOCATIONS:
Locations (16):
- South Korea (16):
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chonnam National University Bitgoeul Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Chungnam National University Hospital, Sejong
  - CHA University Bundang Medical Center, Seongnam
  - EWHA Womans University Mokdong Hospital, Seoul
  - Gangnam Severance Hospita, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kyunghee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No